CLINICAL TRIAL: NCT06440577
Title: Decision Neuroscience of Craving
Brief Title: Craving & Decision-Making
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Anna B. Konova, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2018002176; R01DA054201 (NIH)
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Decision Making
Keywords: Craving; Decision Making; Opioid Use Disorder; Dietary Choice
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Pharmaceutical Preparations; Food

STUDY DESIGN:
Intervention Model Description: Men and women with OUD receiving medications for OUD treatment will complete both the Consumer Items Willingness-to-Pay Task and Snack Foods Willingness-to-Pay Task at two separate task sessions. Non-psychiatric community control participants will complete the Snack Foods Willingness-to-Pay Task.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Consumer Items Willingness-to-Pay Task (Experimental): Men and women with OUD receiving medications for OUD treatment will complete a decision-making task during functional magnetic resonance imaging (fMRI) in which they indicate their willingness-to-pay for everyday consumer items that have associations with drug use or not. Interleaved with blocks of the task, participants will briefly observe stimuli that can produce a change in their psychological state and drug craving, via two psychological/behavioral interventions: Audio-visual stimuli (Neutral-Relaxing) and Audio-visual stimuli (Drug).
  Interventions: Behavioral: Audio-visual stimuli (Neutral-Relaxing); Behavioral: Audio-visual stimuli (Drug)
- Snack Foods Willingness-to-Pay Task (Experimental): Men and women with OUD receiving medications for OUD treatment and control participants from the community will complete a decision-making task during functional magnetic resonance imaging (fMRI) in which they indicate their willingness-to-pay for snack food items that vary in their features (savory, sweet, etc.). Interleaved with blocks of the task, participants will briefly observe stimuli that can produce a change in their psychological state and food craving, via two psychological/behavioral interventions: Audio-visual stimuli (Non-Food) and Audio-visual stimuli (Food).
  Interventions: Behavioral: Audio-visual stimuli (Non-Food); Behavioral: Audio-visual stimuli (Food)

INTERVENTIONS:
Behavioral: Audio-visual stimuli (Neutral-Relaxing) — Audio instruction for participant to allow themselves to experience their feelings followed by 3-min passive viewing of images of neutral everyday objects (e.g., tools, dirt) and their use (construction, gardening).
  Arms: Consumer Items Willingness-to-Pay Task
Behavioral: Audio-visual stimuli (Drug) — Audio instruction for participant to allow themselves to experience their feelings followed by 3-min passive viewing of images of drug paraphernalia (e.g., syringe, tourniquet, heroin) and preparation.
  Arms: Consumer Items Willingness-to-Pay Task
Behavioral: Audio-visual stimuli (Non-Food) — Audio instruction for participant to focus their attention on the experimenter followed by 3-min audio-guided viewing of the experimenter opening/unwrapping an everyday object (e.g., box of crayons) and taking out its contents.
  Arms: Snack Foods Willingness-to-Pay Task
Behavioral: Audio-visual stimuli (Food) — Audio instruction for participant to focus their attention on the experimenter followed by 3-min audio-guided viewing of the experimenter opening/unwrapping a snack (e.g., chocolate bar, bag of chips) and taking out its contents.
  Arms: Snack Foods Willingness-to-Pay Task

SUMMARY:
Craving is the strong desire for something, such as for substances in drug addiction and food or other activities in everyday life. Recent work suggests craving can influence how people make decisions and assign value to choice options available to them, yet the neural mechanisms underlying these interactions between craving and valuation remain unknown. To address this, this study uses cognitive decision-making tasks that measure how much individuals will pay (from a study endowment) to have everyday consumer items or snack foods when they crave something specific (opioids or a specific snack, respectively). First, the study will identify the neural mechanisms for how drug craving (craving for opioids) interacts with valuation for consumer items that have associations with drug use or not in people receiving treatment for opioid use disorder (OUD). This will be evaluated in the activity patterns and interactions among brain regions involved in craving and value assignment during decision-making. Then, the study will examine for parallel mechanisms for how food craving (craving for a specific snack) interacts with valuation for snack food items that have similar features to the craved snack or not in people receiving treatment for OUD and non-psychiatric community control participants.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Willingness to follow study requirements, as evidenced by an ability to provide written informed consent and read, understand, and complete the study procedures
* Minimum of 6th grade reading level

Additional inclusion criteria for participants with OUD:

* Primary diagnosis of OUD encompassing heroin and/or painkiller use
* Receiving medications for OUD treatment on an outpatient basis
* At least 12-month history of opioid use

Exclusion Criteria:

* Unable to speak or read English
* Active psychosis or mania
* Current or past schizophrenia diagnosis
* History of intellectual disability or developmental or neurological disorder, seizures or epilepsy, or loss consciousness lasting more than 30 minutes
* Severe medical conditions requiring hospitalization or that, in the opinion of the study staff could compromise study participation
* MRI contraindications (claustrophobia, nonremovable piercings, certain metal in the body etc.) or pregnancy

Additional exclusion criteria for community control participants:

* Positive urine drug screen
* Current or past problematic substance use other than nicotine, and alcohol abuse confined to college or military service
* Current or past bipolar disorder diagnosis
* Use of central nervous system medications within the past 6 weeks (e.g., antidepressants, Ritalin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Willingness-to-pay | during the task
  The amount that a participant would be willing to pay for different available choice options. This is measured during the decision-making tasks in which participants are shown images of consumer items or snack foods and report how much they would be willing to pay to have the different items in that moment.
fMRI-BOLD activity measured during willingness-to-pay decisions | during the task
  Functional MRI data will be analyzed to measure changes in blood-oxygen-level-dependent (BOLD) signal in specific regions of interest based on prior research (ventral striatum, ventromedial prefrontal cortex, amygdala, and insula) as participants make willingness-to-pay decisions during each task.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Konova, PhD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Rutgers, The State University of New Jersey, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No